CLINICAL TRIAL: NCT02393768
Title: Epigenetic Reprogramming of Monocytes in Patients With Coronary Atherosclerosis
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Canisius-Wilhelmina Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SB EpiCard
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients: patients with documented atherosclerosis on a CCTA
- controls: patients without atherosclerosis on a CCTA

SUMMARY:
In this study, the investigators will determine whether patients with documented atherosclerosis are characterized by specific epigenetic changes in circulating cells of the innate immune system, compared to patients without atherosclerosis.

DETAILED DESCRIPTION:
Rationale: The innate immune system plays a pivotal role in the development and progression of atherosclerosis. Recently, it was reported that monocytes can develop a long-lasting immunological memory after stimulation with various microorganisms, which has been termed 'trained innate immunity'. This memory is induced by epigenetic reprogramming. We hypothesize that trained monocytes augment atherogenesis.

Objective: The main objective is to study whether patients with coronary atherosclerosis show specific epigenetic changes in the promoter regions of pro-inflammatory cytokines and chemokines and whether this correlates with the inflammatory phenotype of these cells.

Study design: Observational study

Study population: Adult patients who have had computed tomography coronary angiography because of chest pain: 20 patients without atherosclerosis and 20 patients with severe atherosclerosis will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male/female),
* aged >18 years,
* admitted to the acute coronary unit of the CWZ hospital for evaluation of chest pain.
* No coronary atherosclerosis
* Or Severe atherosclerosis

Exclusion Criteria:

* Signs or symptoms of a current infection (fever, chills)
* Auto-immune diseases (such as rheumatoid arthritis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients >18 years who have underwent CCTa scanning beacuse of chest pain.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Epigenetic modifications in circulating monocytes | baseline

SECONDARY OUTCOMES:
Inflammatory phenotype | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands